CLINICAL TRIAL: NCT03953690
Title: Acceptability and Persistence of the Use of a Patient-centred E-health Tool for Lupus Patients Followed in a Specialised Centre in France
Acronym: e-LUPUS
Status: Terminated | Type: Observational
Why Stopped: lack of support from doctors and patients
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: DEVILLIERS 2018
Record Dates: First submitted 2019-05-15; First posted 2019-05-16 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Lupus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: use of e-Health service — use of the e-Health e-Lupus account (at least) once a month and encouraged to advise his doctor to consult the entered data before the following consultation

SUMMARY:
Systemic lupus erythematosus (SLE) is a complex disease whose evaluation in daily practice and clinical research requires consideration of several aspects, in particular disease activity and quality of life.

Health systems are increasingly using Patient Reported Outcome measures (PRO) data to measure different dimensions of the disease and its experience.

In addition, there is a growing number of "e-health" tools for patients. Indeed, the collection of health-related data via an electronic system makes it possible to modernise and facilitate communication between patients and doctors within the framework of medical follow-up and therapeutic education. Nevertheless, very few studies measure the acceptability and effective long-term use of such tools, particularly in the context of SLE.

The Sanoïa patient platform is a digital tool already used in therapeutic areas similar to SLE (discoid lupus erythematosus and rheumatoid arthritis), offering a guarantee of safety and a reduced individual cost.

The availability of this health-related quality of life data collection tool via a site and a mobile application adapted to patients with SLE should:

* Facilitate the collection by patients of their quality of life as part of their routine follow-up (patient access)
* Limit the impact of patients' clinical profiles on the frequency of the collection of quality of life data
* Enable internal medicine specialists to systematically use their patients' quality of life data during consultation (physician access).

This study therefore proposes to evaluate this digital platform within the framework of SLE by measuring the distribution of access by physicians according to the data reported by patients and according to the characteristics of the facilities where the subjects were recruited for the study. These data will allow us to evaluate the influence of factors extrinsic to patients on the adoption of the tool. This area has been very poorly evaluated in the few studies that have focused on the adoption of such tools.

ELIGIBILITY:
Inclusion Criteria:

* Adult > 18 years old
* Having given oral consent for participation
* Confirmed systemic lupus diagnosis (ACR criteria)
* Regular follow-up in the centre for more than 12 months
* With Internet access at home
* Affiliated with national health insurance system or other system

Exclusion Criteria:

* Persons subject to a legal protection measure (curatorship, guardianship)
* Persons subject to limited judicial protection
* Adults who are incapable or unable to express their consent
* Patients who cannot read French
* Patients whose cognitive status does not allow them to track their health data on a digital platform
* Patients to be followed up in another centre within 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients attending a consultation in their usual treatment centre
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2020-03-19 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
utilization rate of online patient account | Through study completion, an average of 24 months
  rate of use of the patient account at least twice, at least 1 month apart, over a 12-month period

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire, Dijon, France